CLINICAL TRIAL: NCT04934059
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety of Yuxuebi Tablet in Treating Night Pain of Ankylosing Spondylitis.
Brief Title: Efficacy and Safety of Yuxuebi Tablet in Treating Night Pain of Ankylosing Spondylitis (AS).
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Resources Sanjiu Medical & Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020005P8A02
Record Dates: First submitted 2021-06-08; First posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yuxuebi tablet (Experimental): take 5 tablets once, 3 times a day, for 42（±3）days.
  Interventions: Drug: Yuxuebi tablet
- Placebo tablet (Placebo Comparator): take 5 tablets once, 3 times a day, for 42（±3）days.
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: Yuxuebi tablet — 0.5g/ tablet
  Arms: Yuxuebi tablet
Drug: Placebo tablet — 0.5g/ tablet
  Arms: Placebo tablet

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled clinical trial to evaluate the efficacy and safety of Yuxuebi tablet in treating night pain of Ankylosing Spondylitis.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-65, male or female
2. Confirmed diagnosis of Ankylosing Spondylitis
3. Syndrome of traditional Chinese medicine is blood stasis syndrome
4. ASDAS-CRP (Ankylosing Spondylitis Disease Activity Score)≥2.1
5. Visual analogue scale (VAS) for night pain≥4分
6. Maintained stable doses of Sulfasalazine, Methotrexate, Leflunomide, etc. for more than 1 month if treating with Slow-Acting Antirheumatic Drugs
7. Maintained stable doses of biologics for more than 3 month if treating with biologics
8. Not use Nonsteroidal Antiinflammatory Drugs within 2 weeks
9. Patients who have not participated in other clinical trials within 4 weeks
10. Written informed consent

Exclusion Criteria:

1. Pregnant or breastfeeding or who expecting to conceive
2. Psoriatic arthritis or Enteropathic arthritis
3. AS with iritis or uveitis
4. Abnormal liver function
5. Abnormal kidney function，high level of Creatinine
6. WBC (White Blood Cell)<3.0×10^9/L or with Hematological Disease
7. Patients with poor control of hypertension or diabetes
8. Acute or chronic infectious diseases
9. Severe arrhythmia
10. Patients with malignant tumors or with a history of malignant tumors
11. Drug allergy
12. Patients who had taken Yuxuebi tablet for more than 4 weeks with poor outcome
13. Patients who are treating with Traditional Chinese medicine for promoting blood circulation and removing blood stasis
14. Alcohol or drug abuse
15. Participants who are not suitable for clinical trial under doctors' consideration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Visual analogue scale (VAS) for night pain | Baseline, at day 7, day 14, day 28, day 42 during treatment

SECONDARY OUTCOMES:
Visual analogue scale (VAS) for whole day | Baseline, at day 7, day 14, day 28, day 42 during treatment
BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) | Baseline, at day 28, day 42 during treatment
BASFI (Bath Ankylosing Spondylitis Functional Index) | Baseline, at day 28, day 42 during treatment
BASMI (Bath Ankylosing Spondylitis Metrology Index) | Baseline, at day 28, day 42 during treatment
Syndrome score of traditional Chinese medicine | Baseline, at day 28, day 42 during treatment
  The Evaluation Scale of Syndrome score ranges from 0 (best score) to 15 (worst score).
SF-36 (The Medical Outcomes Study 36-item short-form health survey) | Baseline, at day 42 during treatment
ESR (Erythrocyte Sedimentation Rate) | Baseline, at day 14, day 28, day 42 during treatment
CRP (C-Reactive Protein) | Baseline, at day 14, day 28, day 42 during treatment

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Guang'anmen Hospital, Beijing
  - The First People's Hospital of Guangzhou, Guangzhou
  - The First People's Hospital of Jinzhong, Jinzhong
  - Nanchong Central Hospital, Nanchong
  - Shenzhen Traditional Chinese Medicine Hospital, Shenzhen

IPD SHARING:
Plan to Share IPD: No